CLINICAL TRIAL: NCT03738566
Title: Outcomes of Esophageal Self Dilation for Benign Refractory Esophageal Stricture Management: Randomized Controlled Trial
Brief Title: Outcomes of Esophageal Self Dilation for Benign Refractory Esophageal Stricture Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-000246
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Dilation; Refractory Benign Esophageal Stricture

STUDY DESIGN:
Intervention Model Description: Subjects who agreed to participate in the randomized trial were randomized to standard clinical care consisting of endoscopic dilation as needed versus esophageal self-dilation therapy in a 1:1 ratio using a block randomization approach. Subjects randomized to the standard clinical care group were offered cross-over to the esophageal self-dilation therapy if they failed stand of care. Subjects who agreed to take part in in the observational prospective study either commenced ESDT or continued standard clinical care based on shared decision making with their esophageal provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Standard Clinical Care Endoscopic Dilation Group (Active Comparator): Following standard clinical care consisting of serial endoscopic dilation to achieve an esophageal diameter of at least 10 mm, subjects will undergo repeat upper endoscopy with dilation as needed if their dysphagia relapses which is the current standard of care. A relapse will be considered if a patient developed solid food dysphagia at least once a week.
  Interventions: Procedure: Endoscopic therapy with esophageal dilation
- Esophageal Self-Dilation Therapy (ESDT) Group (Active Comparator): Following standard clinical care consisting of serial endoscopic dilation to achieve an esophageal diameter of at least 10 mm, subjects are instructed to perform esophageal self-dilation twice a day. If dysphagia is adequately controlled, and there was no resistance with passing the dilator, patients will be asked to decrease the frequency of ESDT to daily, weekly, and monthly over an average period of 6 months.
  Interventions: Device: Esophageal self-dilation therapy
- Observational Study Group (Other): Subjects undergo either esophageal self-dilation therapy or continued standard of clinical care base on shared decision making with their esophageal provider.
  Interventions: Device: Esophageal self-dilation therapy; Procedure: Endoscopic therapy with esophageal dilation
- Standard Clinical Care Endoscopic Dilation, Then ESDT (Experimental): Subjects that received standard of clinical care endoscopic dilation who required two endoscopic dilations within 3 months of randomization were considered to have failed standard care and offered cross-over to the self-dilation therapy.
  Interventions: Device: Esophageal self-dilation therapy; Procedure: Endoscopic therapy with esophageal dilation

INTERVENTIONS:
Device: Esophageal self-dilation therapy — Patient learns to pass a polyvinyl dilator orally on a routine basis. Teaching will take over 1-3 training sessions by one of two esophageal physicians and a nurse. Patients will be instructed to start Esophageal self dilation therapy twice a day for at least one week.
  Other Names: ESDT
  Arms: Esophageal Self-Dilation Therapy (ESDT) Group; Observational Study Group; Standard Clinical Care Endoscopic Dilation, Then ESDT
Procedure: Endoscopic therapy with esophageal dilation — A long, flexible tube is inserted down the throat into the esophagus and the narrow area of the esophagus is dilated, or stretched.
  Arms: Observational Study Group; Standard Clinical Care Endoscopic Dilation Group; Standard Clinical Care Endoscopic Dilation, Then ESDT

SUMMARY:
This study is being done to see which treatment is more effective in improving the difficulty of swallowing. Researchers are comparing self-dilation to endoscopic dilation.

DETAILED DESCRIPTION:
Benign esophageal strictures can be challenging condition to treat. The mainstay of treatment is endoscopic dilations. However, 30 to 40% of these strictures recur despite rigorous dilations. Although a consensus definition does not exist, a stricture is typically termed as a refractory benign esophageal stricture (RBES), when there is a failure to maintain luminal patency after at least 5 endoscopic dilations.

Patients with RBES are extremely difficult to manage and the current armamentarium includes repeated endoscopic dilations, corticosteroid or mitomycin C injections, incisional therapy, and/ or temporary stent placement. These procedures are costly, their efficacy can be short-lived, and are associated with great burden both for the patient and clinician.

Esophageal self -dilation therapy (ESDT) is where the patient learns to pass a polyvinyl dilator orally on a routine basis. In past, smaller studies, ESDT appears to be effective for RBES, reducing the number of endoscopic dilations from an average of 21.7 to an average of 1.

ELIGIBILITY:
Inclusion Criteria:

* Refractory benign esophageal stricture defined as an esophageal stricture with persistent dysphagia despite undergoing 5 endoscopic dilations within a 1 year period. Persistent dysphagia will be considered if patients has solid food dysphagia at least once a week

Exclusion Criteria:

* Patient with malignant esophageal stricture
* Angulated stricture which prevents safe passage of Maloney dilator in office setting
* In ability to achieve an esophageal diameter of 10 mm with endoscopic dilation
* Known significant esophageal motor disorder (i.e. achalasia, aperistalsis, functional obstruction, jackhammer, distal esophageal spasm)*
* The presence of esophageal stent
* Inability to learn self-dilation secondary to blindness or cognitive dysfunction
* Use of chronic anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spechler SJ. American gastroenterological association medical position statement on treatment of patients with dysphagia caused by benign disorders of the distal esophagus. Gastroenterology. 1999 Jul;117(1):229-33. doi: 10.1016/s0016-5085(99)70572-x. PMID 10381932
- [Background] Mendelson AH, Small AJ, Agarwalla A, Scott FI, Kochman ML. Esophageal anastomotic strictures: outcomes of endoscopic dilation, risk of recurrence and refractory stenosis, and effect of foreign body removal. Clin Gastroenterol Hepatol. 2015 Feb;13(2):263-271.e1. doi: 10.1016/j.cgh.2014.07.010. Epub 2014 Jul 11. PMID 25019695
- [Background] de Wijkerslooth LR, Vleggaar FP, Siersema PD. Endoscopic management of difficult or recurrent esophageal strictures. Am J Gastroenterol. 2011 Dec;106(12):2080-91; quiz 2092. doi: 10.1038/ajg.2011.348. Epub 2011 Oct 18. PMID 22008891
- [Background] Kochman ML, McClave SA, Boyce HW. The refractory and the recurrent esophageal stricture: a definition. Gastrointest Endosc. 2005 Sep;62(3):474-5. doi: 10.1016/j.gie.2005.04.050. No abstract available. PMID 16111985
- [Background] Hordijk ML, Siersema PD, Tilanus HW, Kuipers EJ. Electrocautery therapy for refractory anastomotic strictures of the esophagus. Gastrointest Endosc. 2006 Jan;63(1):157-63. doi: 10.1016/j.gie.2005.06.016. PMID 16377340
- [Background] Ramage JI Jr, Rumalla A, Baron TH, Pochron NL, Zinsmeister AR, Murray JA, Norton ID, Diehl N, Romero Y. A prospective, randomized, double-blind, placebo-controlled trial of endoscopic steroid injection therapy for recalcitrant esophageal peptic strictures. Am J Gastroenterol. 2005 Nov;100(11):2419-25. doi: 10.1111/j.1572-0241.2005.00331.x. PMID 16279894
- [Background] Eloubeidi MA, Lopes TL. Novel removable internally fully covered self-expanding metal esophageal stent: feasibility, technique of removal, and tissue response in humans. Am J Gastroenterol. 2009 Jun;104(6):1374-81. doi: 10.1038/ajg.2009.133. Epub 2009 Apr 28. PMID 19491851
- [Background] Repici A, Hassan C, Sharma P, Conio M, Siersema P. Systematic review: the role of self-expanding plastic stents for benign oesophageal strictures. Aliment Pharmacol Ther. 2010 Jun;31(12):1268-75. doi: 10.1111/j.1365-2036.2010.04301.x. Epub 2010 Mar 17. PMID 20236257
- [Background] Repici A, Vleggaar FP, Hassan C, van Boeckel PG, Romeo F, Pagano N, Malesci A, Siersema PD. Efficacy and safety of biodegradable stents for refractory benign esophageal strictures: the BEST (Biodegradable Esophageal Stent) study. Gastrointest Endosc. 2010 Nov;72(5):927-34. doi: 10.1016/j.gie.2010.07.031. PMID 21034894
- [Background] Nijhawan S, Udawat HP, Nagar P. Aggressive bougie dilatation and intralesional steroids is effective in refractory benign esophageal strictures secondary to corrosive ingestion. Dis Esophagus. 2016 Nov;29(8):1027-1031. doi: 10.1111/dote.12438. Epub 2015 Nov 6. PMID 26542391
- [Background] Repici A, Small AJ, Mendelson A, Jovani M, Correale L, Hassan C, Ridola L, Anderloni A, Ferrara EC, Kochman ML. Natural history and management of refractory benign esophageal strictures. Gastrointest Endosc. 2016 Aug;84(2):222-8. doi: 10.1016/j.gie.2016.01.053. Epub 2016 Jan 30. PMID 26828759
- [Background] Dzeletovic I, Fleischer DE, Crowell MD, Pannala R, Harris LA, Ramirez FC, Burdick GE, Rentz LA, Spratley RV Jr, Helling SD, Alexander JA. Self-dilation as a treatment for resistant, benign esophageal strictures. Dig Dis Sci. 2013 Nov;58(11):3218-23. doi: 10.1007/s10620-013-2822-7. Epub 2013 Aug 8. PMID 23925823
- [Background] Zehetner J, DeMeester SR, Ayazi S, Demeester TR. Home self-dilatation for esophageal strictures. Dis Esophagus. 2014 Jan;27(1):1-4. doi: 10.1111/dote.12030. Epub 2013 Feb 6. PMID 23387392
- [Background] Kachaamy T, Lott D, Crujido LR, Rentz L, Fleischer D. Esophageal luminal restoration for a patient with a long lye-induced stricture via tunnel endoscopic therapy during a rendezvous procedure followed by self-dilation (with video). Gastrointest Endosc. 2014 Jul;80(1):192-4. doi: 10.1016/j.gie.2014.02.026. No abstract available. PMID 24950654
- [Background] Dzeletovic I, Fleischer DE. Self-dilation for resistant, benign esophageal strictures. Am J Gastroenterol. 2010 Oct;105(10):2142-3. doi: 10.1038/ajg.2010.212. No abstract available. PMID 20927061
- [Background] Dzeletovic I, Fleischer DE, Crowell MD, Kim HJ, Harris LA, Burdick GE, McLaughlin RR, Spratley RV Jr, Sharma VK. Self dilation as a treatment for resistant benign esophageal strictures: outcome, technique, and quality of life assessment. Dig Dis Sci. 2011 Feb;56(2):435-40. doi: 10.1007/s10620-010-1503-z. Epub 2011 Jan 8. PMID 21221805
- [Background] Lee HJ, Lee JH, Seo JM, Lee SK, Choe YH. A single center experience of self-bougienage on stricture recurrence after surgery for corrosive esophageal strictures in children. Yonsei Med J. 2010 Mar;51(2):202-5. doi: 10.3349/ymj.2010.51.2.202. Epub 2010 Feb 12. PMID 20191010
- [Background] Wong KK, Hendel D. Self-dilation for refractory oesophageal strictures: an Auckland City Hospital study. N Z Med J. 2010 Aug 27;123(1321):49-53. PMID 20927157
- [Background] Bapat RD, Bakhshi GD, Kantharia CV, Shirodkar SS, Iyer AP, Ranka S. Self-bougienage: long-term relief of corrosive esophageal strictures. Indian J Gastroenterol. 2001 Sep-Oct;20(5):180-2. PMID 11676328
- [Derived] Halland M, Prichard DO, Kahn A, Lavey CJ, Katzka DA, Alexander JA. Esophageal Self-Dilation in Benign Refractory Esophageal Strictures: Outcomes from a Randomized Controlled Trial and a Prospective Observational Study. Dig Dis Sci. 2024 Aug;69(8):2883-2889. doi: 10.1007/s10620-024-08402-z. Epub 2024 May 29. PMID 38811502
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 subjects randomized to self-dilation group and 6 subjects randomized to standard of care with repeat endoscopy and dilations as needed at symptoms recurrence. 5 subjects from the standard of care group crossed over to receive self-dilation because they were considered treatment failures due to requiring 2 endoscopic dilation after 3 months of study participation. 14 subjects choose not to participate in the randomized trial, but did agree to be followed in a prospective observational group.
Period: Initial Study Phase
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
Started | 6 | 6 | 14 | 0
Completed | 0 | 4 | 12 | 0
Not Completed | 6 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Treatment failure | 5 | 0 | 0 | 0
Period: Cross-over for Treatment Failure
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
Started | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 26 participants were enrolled in the overall study. 5 subjects in the Standard Clinical Care Endoscopic Dilation Group were considered treatment failures and were crossed over to the self-dilation group, resulting in a total of 31 participants analyzed for the Baseline Measures overall.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT | Total
Number analyzed (Participants) | 6 | 6 | 14 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Data collected from the cross over study group are being reported separately to avoid multi-counted participants. Population: Data are reported separately for the initial phase and cross over phase. Data was not collected in the initial study phase for the Standard Clinical Care Endoscopic Dilation, Then ESDT group. Data was not collected in the cross-over for Treatment Failure phase for Standard Clinical Care Endoscopic Dilation Group, Esophageal Self-Dilation Therapy (ESDT) Group, or Observational Study Group as these groups were only part of the initial study phase.
  years
    Initial Study Phase: number analyzed (Participants) | 6 | 6 | 14 | 0 | 26
    Initial Study Phase | 64.0 (11.0) | 62.3 (9.6) | 62 (15) |  | 62.9 (12.3)
    Cross-over for Treatment Failure: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Cross-over for Treatment Failure |  |  |  | 65 (7) | 65 (7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected from the cross over study group are being reported separately to avoid multi-counted participants.
  Participants
    Initial Study Phase: number analyzed (Participants) | 6 | 6 | 14 | 0 | 26
    Initial Study Phase: Female | 3 | 4 | 7 | 0 | 14
    Initial Study Phase: Male | 3 | 2 | 7 | 0 | 12
    Cross-over for Treatment Failure: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    Cross-over for Treatment Failure: Female | 0 | 0 | 0 | 3 | 3
    Cross-over for Treatment Failure: Male | 0 | 0 | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Initial Study Phase Population: Data collected from the cross over study group are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 6 | 6 | 14 | 0 | 26
    United States | 6 | 6 | 14 |  | 26
Region of Enrollment [Number; unit: participants] — Cross-over for Treatment Failure Population: Data collected from the cross over study group are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
    United States |  |  |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Endoscopic Interventions
Description: Number of endoscopies required in a 6 month interval in subjects who achieved at least a 10-12 mm esophageal diameter during serial dilation for refractory benign esophageal stricture (RBES) and were subsequently treated with ESDT versus standard clinical care
Time Frame: 6 months following serial dilation
Measure: Number; unit: endoscopies
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
Number analyzed (Participants) | 5 | 6 | 14 | 4
endoscopies | 12 | 11 | 12 | 7

2. Secondary Outcome: Length of Days Intervention Free
Description: Number of days from start of study participation to 1st endoscopic intervention for recurrent dysphagia
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group
Number analyzed (Participants) | 5 | 6 | 14
days | 7 [2 to 33] | 82 [39 to 124] | 147 [113.5 to 166.5]

3. Secondary Outcome: Mayo Dysphagia Questionnaire (MDQ-30) at Baseline
Description: The MDQ-30 provides a series of questions for patients regarding their swallowing difficulties over the past 30 days. Participants were asked to rate the severity of their troubles swallowing on a scale of 0 to 10; 0 being "Not at all severe" and 10 being "Very severe"
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group
Number analyzed (Participants) | 6 | 6 | 14
score on a scale | 7.16 (1.16) | 7.56 (1.44) | 5.36 (2.17)

4. Secondary Outcome: Mayo Dysphagia Questionnaire (MDQ-30) at 12 Months
Description: as for outcome 3
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
Number analyzed (Participants) | 4 | 12 | 4
score on a scale | 5.55 (2.07) | 5.83 (3.60) | 5.17 (2.04)

5. Secondary Outcome: Clinically Significant Adverse Events
Description: Number of clinically significant adverse events including perforation, bleeding and pain
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
Number analyzed (Participants) | 6 | 6 | 14 | 5
events | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 12 months on all participants.
Arm/Group | Standard Clinical Care Endoscopic Dilation Group | Esophageal Self-Dilation Therapy (ESDT) Group | Observational Study Group | Standard Clinical Care Endoscopic Dilation, Then ESDT
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/14 | 1/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/14 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Clinical Care Endoscopic Dilation Group (N=6) | Esophageal Self-Dilation Therapy (ESDT) Group (N=6) | Observational Study Group (N=14) | Standard Clinical Care Endoscopic Dilation, Then ESDT (N=5)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03738566/Prot_SAP_000.pdf